CLINICAL TRIAL: NCT05067062
Title: Effects of Intake Duration of New Zealand Blackcurrant Extract on Physiological, Cardiovascular and Metabolic Responses at Rest and During Moderate-intensity Exercise in Healthy Males
Brief Title: Intake Duration Effects of Blackcurrant on Cardiovascular and Metabolic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chichester (Other)
Responsible Party: Principal Investigator, Mark Eilisabeth Willems, Professor of Exercise Physiology, University of Chichester
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MW1718NZBCduration
Record Dates: First submitted 2021-09-10; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: no Conditions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new zealand blackcurrant extract (Active Comparator): Capsules will be take daily or every other day.
  Interventions: Dietary Supplement: New Zealand blackcurrant extract
- control (Placebo Comparator): no capsules will be provided.
  Interventions: Dietary Supplement: New Zealand blackcurrant extract

INTERVENTIONS:
Dietary Supplement: New Zealand blackcurrant extract — Capsules taken daily or intermittent

SUMMARY:
Study will examine the metabolic, physiological and cardiovascular changes by intake of New Zealand blackcurrant extract at rest and during moderate-intensity treadmill walking in healthy males.

DETAILED DESCRIPTION:
The investigators will examine effects of acute intake, intermittent intake and chronic intake of New Zealand blackcurrant extract using indirect calorimetry and hemodynamic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smokers
* Not taking any supplements
* No known allergy to berries or berry products

Exclusion Criteria

* Sedentary
* Known high blood pressure
* Smoking
* On medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in heart rate from baseline with acute intake, one week and two weeks intake of New Zealand blackcurrant extract | baseline, acute, one week and two weeks
  The investigators will use a beat-to-beat blood pressure monitoring system (Portapres® Model 2, Finapres Medical Systems BV, Amsterdam, The Netherlands). The Portapres® is a beat-to-beat finger pressure analyser that allows the non-invasive continuous measurement of hemodynamic parameters. The finger cuff will be positioned around the same finger of the left hand for each testing. All measurements will be taken in rest and during moderate-intensity exercise.
  Heart rate will be measured in beats/min.
Changes in stroke volume from baseline with acute intake, one week and two weeks intake of New Zealand blackcurrant extract | baseline, acute, one week and two weeks
  The investigators will use a beat-to-beat blood pressure monitoring system (Portapres® Model 2, Finapres Medical Systems BV, Amsterdam, The Netherlands). The Portapres® is a beat-to-beat finger pressure analyser that allows the non-invasive continuous measurement of hemodynamic parameters. The finger cuff will be positioned around the same finger of the left hand for each testing. All measurements will be taken in rest and during moderate-intensity exercise.
  Stroke volume will be measured in mL.
Changes in cardiac output from baseline with acute intake, one week and two weeks intake of New Zealand blackcurrant extract | baseline, acute, one week and two weeks
  The investigators will use a beat-to-beat blood pressure monitoring system (Portapres® Model 2, Finapres Medical Systems BV, Amsterdam, The Netherlands). The Portapres® is a beat-to-beat finger pressure analyser that allows the non-invasive continuous measurement of hemodynamic parameters. The finger cuff will be positioned around the same finger of the left hand for each testing. All measurements will be taken in rest and during moderate-intensity exercise.
  Cardiac output will be measured in L/min.
Changes in blood pressure from baseline with acute intake, one week and two weeks intake of New Zealand blackcurrant extract | baseline, acute, one week and two weeks
  The investigators will use a beat-to-beat blood pressure monitoring system (Portapres® Model 2, Finapres Medical Systems BV, Amsterdam, The Netherlands). The Portapres® is a beat-to-beat finger pressure analyser that allows the non-invasive continuous measurement of hemodynamic parameters. The finger cuff will be positioned around the same finger of the left hand for each testing. All measurements will be taken in rest and during moderate-intensity exercise.
  Systolic, diastolic and mean arterial blood pressure will be measured in mmHg.
Changes in total peripheral resistance from baseline with acute intake, one week and two weeks intake of New Zealand blackcurrant extract | baseline, acute, one week and two weeks
  The investigators will use a beat-to-beat blood pressure monitoring system (Portapres® Model 2, Finapres Medical Systems BV, Amsterdam, The Netherlands). The Portapres® is a beat-to-beat finger pressure analyser that allows the non-invasive continuous measurement of hemodynamic parameters. The finger cuff will be positioned around the same finger of the left hand for each testing. All measurements will be taken in rest and during moderate-intensity exercise.
  Total peripheral resistance will be measured in (mmHg·min)/L

SECONDARY OUTCOMES:
Changes in oxygen consumption from baseline with acute intake, one week and two weeks intake. | baseline, acute, one week and two weeks
  The investigators will use Douglas bags to collect expired air. Indirect calorimetry techniques will be used to measured oxygen consumption and carbon dioxide production and allow quantification of carbohydrate and fat oxidation in rest and during moderate-intensity treadmill walking.
  Oxygen consumption will be measured in L/min
Changes in carbon dioxide production from baseline with acute intake, one week and two weeks intake. | baseline, acute, one week and two weeks
  The investigators will use Douglas bags to collect expired air. Indirect calorimetry techniques will be used to measured oxygen consumption and carbon dioxide production and allow quantification of carbohydrate and fat oxidation in rest and during moderate-intensity treadmill walking.
  Carbon dioxide production will be measured in L/min.
Changes in respiratory exchange ratio from baseline with acute intake, one week and two weeks intake. | baseline, acute, one week and two weeks
  The investigators will use Douglas bags to collect expired air. Indirect calorimetry techniques will be used to measured oxygen consumption and carbon dioxide production and allow quantification of carbohydrate and fat oxidation in rest and during moderate-intensity treadmill walking.
  Respiratory exchange ratio is unitless and calculated from the ratio of carbon dioxide production and oxygen consumption.
Changes in carbohydrate oxidation from baseline with acute intake, one week and two weeks intake. | baseline, acute, one week and two weeks
  The investigators will use Douglas bags to collect expired air. Indirect calorimetry techniques will be used to measured oxygen consumption and carbon dioxide production and allow quantification of carbohydrate and fat oxidation in rest and during moderate-intensity treadmill walking.
  Carbohydrate oxidation is calculated using carbon dioxide production and oxygen consumption and expressed in g/min.
Changes in fat oxidation from baseline with acute intake, one week and two weeks intake. | baseline, acute, one week and two weeks
  The investigators will use Douglas bags to collect expired air. Indirect calorimetry techniques will be used to measured oxygen consumption and carbon dioxide production and allow quantification of carbohydrate and fat oxidation in rest and during moderate-intensity treadmill walking.
  Fat oxidation is calculated using carbon dioxide production and oxygen consumption and expressed in g/min.

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Willems, PhD, Principal Investigator — University of Chichester
Locations (1):
- Mark Willems, Chichester, West Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No
But will be provide on request.

REFERENCES:
- [Background] Sahin PhD MA, Bilgic PhD P, Montanari MSc S, Willems PhD MET. Intake Duration of Anthocyanin-Rich New Zealand Blackcurrant Extract Affects Metabolic Responses during Moderate Intensity Walking Exercise in Adult Males. J Diet Suppl. 2021;18(4):406-417. doi: 10.1080/19390211.2020.1783421. Epub 2020 Jun 24. PMID 32578472
- [Result] Sahin PhD MA, Bilgic PhD P, Montanari MSc S, Willems PhD MET. Daily and Not Every-Other-Day Intake of Anthocyanin-Rich New Zealand Blackcurrant Extract Alters Substrate Oxidation during Moderate-Intensity Walking in Adult Males. J Diet Suppl. 2022;19(1):49-61. doi: 10.1080/19390211.2020.1841356. Epub 2020 Oct 29. PMID 33118421